CLINICAL TRIAL: NCT00431392
Title: Mechanisms of Choroidal Blood Flow Changes During Dark/Light Transitions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OPHT-180601
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2007-02-05 (Estimated); Status verified 2007-01

CONDITIONS: Regional Blood Flow; Ocular Physiology
Keywords: Choroidal blood flow; NO-synthase; light/dark transition
MeSH Terms: interventions — Phenylephrine; omega-N-Methylarginine; Propranolol; Atropine

INTERVENTIONS:
Drug: Phenylephrine
Drug: NG-Monomethyl-L-Arginine
Drug: Propanolol
Drug: Atropine

SUMMARY:
There is evidence from a variety of animal studies that choroidal blood flow is under neural control. By contrast, only little information is available from human studies. Recent results indicate that a light/dark transition is associated with a short lasting reduction in choroidal blood flow. We have shown that during unilateral dark/light transition both eyes react with choroidal vasoconstriction strongly indicating a neural mechanism.

The present studies investigate this possibility by using pharmacological interventions. The pharmacological agents tested include a nitric oxide synthase inhibitor, an alpha-receptor agonist (as a control substance for the blood pressure increasing nitric oxide synthase inhibitor), a muscarinic receptor blocker, and a non-specific beta-blocker. These drugs were chosen on the basis of previous animal experiments, as the systems, which are specifically influenced by these substances, are likely involved in neural control of choroidal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile (Must et al. 1991)
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2001-09

PRIMARY OUTCOMES:
choroidal blood flow
fundus pulsation amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria